CLINICAL TRIAL: NCT06274086
Title: Safety and Clinical Outcomes of Two-session Catheter-directed Sclerotherapy Using Ethanol for Endometrioma
Brief Title: Two-session Catheter-directed Sclerotherapy Using Ethanol for Endometrioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hoon Shin, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2022-2027-0001
Record Dates: First submitted 2024-02-08; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Sclerotherapy; Endometrioma
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Two-session catheter-directed sclerotherapy (Experimental): Each patient received two sessions of catheter-directed sclerotherapy for endometrioma 1 day apart with the catheter left in situ overnight.
  Interventions: Procedure: Two-session catheter-directed sclerotherapy

INTERVENTIONS:
Procedure: Two-session catheter-directed sclerotherapy — After receiving the first session of catheter-directed sclerotherapy, each patient carries the catheter overnight and is closely monitored in the patient ward. Then, the patient receives the second session the next day. The catheter is removed after the second session.
  The procedure was performed under intravenous sedoanalgesia using a combination of 25 mg pethidine hydrochloride and 50 mg fentanyl. Devices used during the procedure included:
  * An 18-gauge, 20-cm Chiba biopsy needle (Cook, Bloomington, IN, USA);
  * A 0.035-inch hydrophilic guidewire (Terumo, Tokyo, Japan);
  * A 7- or 8.5-F pigtail catheter (Dawson-Mueller Drainage Catheter; Cook).

SUMMARY:
The goal of this clinical trial is to evaluate the safety and clinical outcomes of two-session catheter-directed sclerotherapy (CDS) with 96% ethanol in patients with endometrioma. The main question it aims to answer is:

• Is two-session CDS with 96% ethanol safe and effective for treating endometrioma?

Participants will:

* Receive the first session CDS for endometrioma
* Carry the catheter overnight and be monitored in the patient ward
* Receive the second session CDS the next day

DETAILED DESCRIPTION:
Catheter-directed sclerotherapy has been reported as an effective treatment for endometrioma. However, whether the sclerosing agent should be retained inside the endometrioma was controversial. To increase the contact between the sclerosing agent and the endometrioma wall, two-session catheter-directed sclerotherapy using 96% ethanol was attempted, and safety and clinical outcomes were assessed in patients with endometrioma.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Symptom manifestation as endometriosis (i.e., dysmenorrhea, dyspareunia, and lower abdominal or pelvic pain)
* Endometrioma ≥ 3 cm confirmed on ultrasound
* No evidence of solid lesions on ultrasound
* No suspected extraovarian endometriosis

Exclusion Criteria:

* History of gynecologic malignancy
* Active inflammation or infection
* Abnormal coagulation profile
* Loss to follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Recurrence | Recurrence was assessed at 1, 3, and 6 months after the procedure.
  Recurrence of endometrioma was assessed

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hoon Shin, MD, PhD, Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea